CLINICAL TRIAL: NCT04837716
Title: A Phase 1b Study of Ensartinib in Combination With Platinum-Based Chemotherapy and Bevacizumab in ALK-Positive Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Ensartinib, Carboplatin, Pemetrexed and Bevacizumab for the Treatment of Stage IIIC or IV or Recurrent ALK-Positive Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0838; NCI-2021-02560 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0838 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Carboplatin; ensartinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ensartinib, carboplatin, pemetrexed, bevacizumab) (Experimental): INDUCTION THERAPY: Patients receive ensartinib PO QD on days 1-21, carboplatin IV over 15-60 minutes on day 1, pemetrexed IV over 10 minutes on day 1 and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive ensartinib PO QD on days 1-21 and bevacizumab IV over 30-90 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Drug: Ensartinib; Drug: Pemetrexed

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; Zirabev
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Ensartinib — Given PO
  Other Names: X-396
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy

SUMMARY:
This phase Ib trial finds the best dose and side effects of ensartinib and its effects when given with carboplatin, pemetrexed and bevacizumab for in treating patients with ALK-positive non-small cell lung cancer that is stage IIIC or IV, or has come back (recurrent). Ensartinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as carboplatin and pemetrexed, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bevacizumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Giving ensartinib, carboplatin, pemetrexed and bevacizumab may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of ensartinib in combination with carboplatin, pemetrexed and bevacizumab in patients with ALK-rearranged advanced non-small cell lung cancer (NSCLC).

II. Determine the recommended phase 2 dose (RP2D) of ensartinib in combination with carboplatin, pemetrexed and bevacizumab.

SECONDARY OBJECTIVES:

I. To determine an objective response rate (ORR) in patients with ALK-rearranged advanced NSCLC treated with ensartinib in combination with carboplatin, pemetrexed and bevacizumab using modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

II. To determine progression-free survival (PFS). III. To determine overall survival.

EXPLORATORY OBJECTIVE:

I. To determine biomarkers associated with response and resistance to the study combination.

OUTLINE: This is a dose de-escalation study of ensartinib and fixed-dose carboplatin, pemetrexed, and bevacizumab followed by a dose-expansion study.

INDUCTION THERAPY: Patients receive ensartinib orally (PO) once daily (QD) on days 1-21, carboplatin intravenously (IV) over 15-60 minutes on day 1, pemetrexed IV over 10 minutes on day 1 and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive ensartinib PO QD on days 1-21 and bevacizumab IV over 30-90 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of stage IV (metastatic) or recurrent or stage IIIc NSCLC (recurrent or stage IIIC NSCLC must be not a candidate for definitive multimodality therapy)
* Documented ALK re-arrangement as detected by: (1) fluorescence in situ hybridization (FISH), (2) immunohistochemistry (IHC), (3) tissue next generation sequencing (NGS), or (4) cell free deoxyribonucleic acid (cfDNA) NGS using Clinical Laboratory Improvement Amendments (CLIA) certified laboratory
* Subjects can be enrolled as (1) treatment naive (2) after progression on any number of prior ALK tyrosine kinase inhibitors (TKIs). Prior adjuvant platinum-based chemotherapy and platinum-based chemotherapy for metastatic disease is allowed if completed > 12 months from the study treatment start date with one exception: a patient may be eligible if started on chemotherapy while waiting for ALK testing results, provided no more than two cycles of chemotherapy were administered and no evidence of disease progression
* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Aged at least 18 years
* Brain metastases allowed if asymptomatic at study baseline. Patients must be not on steroids, with the maximum size of brain lesion not exceeding 30 millimeters. If patients have neurological symptoms or signs due to central nervous system (CNS) metastases, patients need to complete whole brain radiation or focal treatment at least 14 days before start of study treatment and be asymptomatic on stable or decreasing doses of corticosteroids at baseline
* Ability to swallow and retain oral medications
* Absolute neutrophil count (ANC) >= 1500/mm^3 /L
* Platelet count >= 100,000/mm^3
* Hemoglobin (Hb) at least 9 g/dL (or 5.69 mmol/L) at baseline
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or creatinine clearance (CrCl) >= 60 mL/minute for subjects with creatinine levels > 1.5 x the institutional ULN
* Serum total bilirubin less than or equal to =< 1.5 x ULN or direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN except for subjects with liver metastases (mets) for whom ALT and AST should be =< 5 x ULN
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated PTT (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy if PT or PTT is within therapeutic range of intended use of anticoagulant
* Female patients of childbearing potential must have a negative pregnancy test documented at time of screening
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to use a highly effective method of contraception from the time of signing the informed consent through 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or
  * Agree to completely abstain from heterosexual intercourse
* Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol

Exclusion Criteria:

* Use of an investigational drug within 21 days prior to the first dose of study drug. Note that to be eligible, any drug-related toxicity should have recovered to grade 2 or less, with the exception of alopecia
* Major surgery within the last 4 weeks or radiotherapy within the last 14 days
* Patients with leptomeningeal disease are ineligible
* Patients with a previous malignancy within the past 2 years (other than curatively treated basal cell carcinoma of the skin, in situ carcinoma of the cervix, or any cancer that is considered to be cured and have no impact on PFS and overall survival [OS] for the current NSCLC)
* Concomitant systemic use of anticancer herbal medications. These should be stopped prior to study entry
* Patients receiving:

  * Strong CYP3A inhibitors (including, but not limited to, atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, grapefruit, grapefruit juice)
  * Strong CYP3A inducers (including, but not limited to, carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, St. John's wort)
  * CYP3A substrates with narrow therapeutic window (including, but not limited to, alfentanil, cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, tacrolimus)
* Women who are pregnant or breastfeeding
* Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of study medications
* Patients at risk for GI perforation
* Clinically significant cardiovascular disease including:

  * Corrected QT per Fridericia's formula (QTcF) interval > 450 ms for men and > 470 ms for women, symptomatic bradycardia < 45 beats per minute or other significant electrocardiogram (ECG) abnormalities in the investigator's opinion
  * Clinically uncontrolled hypertension in the investigator's opinion (e.g., blood pressure > 160/100 mmHg; note that isolated elevated readings considered to not be indicative of uncontrolled hypertension are allowed)
  * The following within 6 months prior to cycle 1 day 1:

    * Congestive heart failure (New York Heart class III or IV)
    * Arrhythmia or conduction abnormality requiring medication. Note: patients with atrial fibrillation/flutter controlled by medication and arrhythmias controlled by pacemakers are eligible
    * Severe/unstable angina, coronary artery/peripheral bypass graft, or myocardial infarction
    * Cerebrovascular accident or transient ischemia
* Patients who are immunosuppressed (including known human immunodeficiency virus [HIV] infection), have a serious active infection at the time of treatment, have interstitial lung disease/pneumonitis, or have any serious underlying medical condition that would impair the ability of the patient to receive protocol treatment. Patients with controlled hepatitis C, in the investigator's opinion, are allowed. Patients with known hepatitis B must be hepatitis B virus e antigen (HBeAg) and HB viral deoxyribonucleic acid (DNA) negative for enrollment. Note that, because of the high prevalence, all patients in the Asia-Pacific region (except Australia, New Zealand, and Japan) must be tested and, if hepatitis B surface antigen (HBsAg) positive, must be HBeAg and HB viral DNA negative for enrollment
* Known hypersensitivity to tartrazine, a dye used in the ensartinib 100 mg capsule
* Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol or would impart excessive risk associated with study participation that would make it inappropriate for the patient to be enrolled
* Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2027-09-23 (Estimated); Study Completion 2027-09-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days
  The toxicity rate will be estimated with their exact 95% confidence intervals.
Recommended phase 2 dose | Up to 21 days
  Will employ the Bayesian optimal interval (BOIN) design (Liu and Yuan, 2015; Yuan et al., 2016) to find the maximum tolerated dose of ensartinib in combination with carboplatin, pemetrexed and bevacizumab.

SECONDARY OUTCOMES:
Objective response rate | Up to 1.5 years
  Assessed using modified Response Evaluation Criteria in Solid Tumors (1.1). The response rate will be estimated with their exact 95% confidence intervals.
Progression-free survival | Up to 1.5 years
  Will be estimated using the method of Kaplan and Meier.
Overall survival | Up to 1.5 years
  Will be estimated using the method of Kaplan and Meier.

OTHER OUTCOMES:
Biomarkers associated with response and resistance | Up to 1.5 years
  The difference in the biomarkers between responders and non-responders will be evaluated by Fisher's exact test for categorical biomarkers or Wilcoxon rank sum test for continuous biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Y Elamin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT04837716/ICF_000.pdf